CLINICAL TRIAL: NCT06785727
Title: StAtins in Frail OldEr Patients with Ischemic Stroke or Transient Ischemic Attack - the Randomized Controlled Trial
Acronym: SAFEST - RCT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. dr. Nathalie van der Velde (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Sponsor-Investigator, Prof. dr. Nathalie van der Velde, Full Professor Geriatric medicine (internal medicine), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-502059-79-00
Record Dates: First submitted 2023-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: statin; ischemic stroke; transient ischemic attack; quality of life
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Fluvastatin; Pravastatin; Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Intervention Model Description: Multicentre prospective randomized open-label approach with blinded end-points evaluation (PROBE)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prescribing a statin (Experimental): Newly prescribing a statin
  Interventions: Drug: Statin (atorvastatin, fluvastatin, pravastatin, rosuvastatin or simvastatin)
- Not prescribing a statin (No Intervention): Not prescribing a statin

INTERVENTIONS:
Drug: Statin (atorvastatin, fluvastatin, pravastatin, rosuvastatin or simvastatin) — The intervention group receives statin treatment following the current "Herseninfarct en Hersenbloeding" guideline. The intensity and target value of statin treatment are determined according to this national guideline. Which statin (atorvastatin, fluvastatin, pravastatin, rosuvastatin, simvastatin) will be selected and what dose will be prescribed is left to the discretion of the treating neurologist. The statins are registered in the Netherlands and use will be according to the licenses of the products. They will be collected at the local pharmacy by the patient (following practice as usual).
  Other Names: Lipitor, Lescol XL, Crestor, Zocor
  Arms: Prescribing a statin

SUMMARY:
Two Dutch guidelines (Stroke and Cardiovascular Risk Management) provide conflicting advice on optimal statin treatment in older patients. In the SAFEST - RCT, the investigators will assess the impact of starting versus not starting a statin in frail individuals aged 70 and above with a recent ischemic stroke or transient ischemic attack (TIA) on their health-related quality of life and Major Adverse Cardiovascular Events (MACE) free survival during a two-year follow-up period.

DETAILED DESCRIPTION:
Objective: To assess the impact of starting versus not starting a statin in frail individuals aged 70 and above with a recent ischemic stroke or transient ischemic attack (TIA) on their health-related quality of life and MACE free survival during a two-year follow-up period.

Study population: The patient population consists of frail older (>=70 yrs) patients with a recent acute ischemic stroke or TIA who are admitted to the hospital or visit the outpatient clinic or emergency department for diagnostic evaluation, and who were not receiving statin treatment at the time of the acute event. Frailty is defined by a pre-event Clinical Frailty Scale (CFS) score of 4-7 and/or a post-event score of 6-7.

Description of intervention(s): Participants in the intervention group will start with a statin with target values following the Dutch stroke guideline. The control group will not start with a statin, aligning with the Dutch Cardiovascular Risk Management (CVRM) guideline recommendations.

Outcome measures:

This study has two co-primary endpoints: (1) Health-Related Quality of Life (HrQoL), using the Patient-Reported Outcomes Measurement Information System - Global-10 (PROMIS-10) and (2) Major Adverse Cardiovascular Events (MACE) free survival, after 2 years. We will evaluate these two co-primary outcomes at multiple time points, specifically at 3, 6, 12, 18, and 24 months. For patients enrolled in the beginning of recruitment, an extended follow-up of three years will be conducted to provide additional insights into the two primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* age = 70 years or older at the time of ischemic stroke or TIA;
* inclusion within 6 weeks after diagnosis of ischemic stroke or TIA;
* not using statin therapy at the time of the index event;
* frailty as defined by a pre-event score of 4-7 and/or post-event score of 6-7 on the validated Clinical Frailty Scfale.[49]

Exclusion Criteria:

* Patients with a stroke or TIA of non-atherosclerotic etiology.
* Previous serious adverse drug reactions (defined as an adverse reaction that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is a birth defect40) to statins or other contraindications to statin use.
* Very severe frailty or very limited life expectancy (< 6 months) as defined by a score >= 8 points on the validated Clinical Frailty Scale.
* Inability to communicate in Dutch.
* Inability to respond to questions, either independently or with the assistance of a proxy (a proxy is allowed to assist by writing on behalf of the participant in cases of physical incapacity or by discussing questions with the participant, but the proxy cannot make decisions for the participant).
* Inability or unwillingness to provide written informed consent, either independently or with the assistance of a proxy (a proxy is allowed to assist by writing on behalf of the participant in cases of physical incapacity or by discussing the consent form with the participant, but the proxy cannot make decisions or provide consent on behalf of the participant).
* Extremely high-risk patients, i.e. patients who have had two or more cardiovascular events within a period of one year.

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HrQoL) | 3, 6, 12, 18, 24 (and 36) months.
  This will be measured using the PROMIS-10 scale scores (ranging from 0 to 100, with higher scores indicating better health), including global mental health and global physical health subscales. Measurements at 3, 6, 12, 18, 24 (and 36) months.
Major Adverse Cardiovascular Events (MACE) free survival | 3, 6, 12, 18, 24 (and 36) months.
  Classical 3-point MACE (cardiovascular death, nonfatal myocardial infarction, or nonfatal stroke) and non-cardiovascular death. Measurements at3, 6, 12, 18, 24 (and 36) months.

SECONDARY OUTCOMES:
Functional Outcome | 1 and 2 years
  This will be assessed using the modified Rankin Scale (mRS) 49, with scores ranging from 0 to 6 (lower scores indicating better function).
Cognition MoCA | 1 and 2 years
  will be measured using the Montreal Cognitive Assessment (MoCA)51 or the Telephone version of the MoCA (T-MOCA)
Number of falls | 1 and 2 years
  Falls, measured using the falls calender. Participant returns the fall calender every 3 months.
Time to first fall | 2 years
  Falls, measured using the falls calender. Participant returns the fall calender every 3 months.
General quality of life EuroQol Questionnaire (EQ-5D-5L) | 1 and 2 years
  General QoL measure by EuroQol Questionnaire (EQ-5D-5L). This will be used to calculate the cost-effectiveness analysis (CAE). Possible scores range from 0-100, the higher, the better.
Societal costs | 1 and 2 years
  Societal costs measured by The Older Persons and Informal Caregivers Survey - Minimum Data Set (TOPICS-MDS) (questions 23 - 37)
Cardiovascular Risk Status | 1 and 2 years
  method of assessing is to be decided.

CONTACTS AND LOCATIONS:
Overall Officials: Renske van den Berg, Prof. dr., Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands; Nathalie van der Velde, Prof. dr., Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The SAFEST database can be requested by other researchers. These requests will be reviewed according the requirements for sharing SAFEST data.
Supporting Information: Study Protocol, SAP
Time Frame: After data-collection/analysis.
Access Criteria: Requirements for sharing SAFEST data include:
  * privacy laws of the Netherlands, policy of NFU and AmsterdamUMC must be followed
  * data will anonymously
  * data can only be used to study the research question for which participants signed the ICF
  * data will not be shared for commercial purposes.

REFERENCES:
- [Derived] Prins SR, Damoiseaux-Volman BA, Vermeer SE, Bossuyt PMM, Van Eekelen R, Bosmans JE, Van Poelgeest EP, Martens FMAC, Emmelot-Vonk MH, Verstraete E, Muller M, Moll Van Charante EP, Lindhout M, Van Der Velde N, Van Den Berg-Vos RM. Rationale and design of 'StAtins in Frail oldEr patients with ischemic Stroke or Transient ischemic attack-the Randomized Controlled Trial' (SAFEST-RCT). BMJ Neurol Open. 2025 Oct 5;7(2):e001297. doi: 10.1136/bmjno-2025-001297. eCollection 2025. PMID 41070271